CLINICAL TRIAL: NCT01420068
Title: A Multicenter, Double-blind 52 to 104 Week Off-therapy Extension Study to Evaluate the Long Term Growth and Development of Pediatric Hypertensive Patients 6 - 17 Years of Age Previously Treated With Aliskiren in Studies CSPP100A2365 and/or CSPP100A2365E1
Brief Title: 52-104 Week Off-therapy Second Extension to Study CSPP100A2365
Status: Completed | Type: Observational
Sponsor: Noden Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: CSPP100A2365E2; 2011-004411-22
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2018-09

CONDITIONS: Hypertension
Keywords: Pediatric; hypertension; aliskiren
MeSH Terms: conditions — Hypertension | interventions — aliskiren

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- All patients: All patients previously treated with study medication in the CSPP100A2365 and CSPP100A2365E1 studies.
  Interventions: Drug: SPP100

INTERVENTIONS:
Drug: SPP100

SUMMARY:
52-104 week off-therapy second extension to study CSPP100A2365 to assess growth and development in pediatric hypertensive patients previously treated with aliskiren in studies SPP100A2365 and SPP100A2365E1

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of study CSPP100A2365E1
* Patients must meet inclusion criteria set forth for trials CSPP100A2365 and CSPP100A2365E1
* Informed consent/ patient assent

Exclusion Criteria:

•Patients who did not successfully complete studies CSPP100A2365 and CSPP100A2365E1

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric hypertensive patients 6 - 17 years of age previously treated with aliskiren in studies CSPP100A2365 and/or CSPP100A2365E1
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2011-08-19 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (10):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Dalton, Georgia
  - Novartis Investigative Site, Lewiston, Idaho
  - Novartis Investigative Site, Hattiesburg, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Amarillo, Texas
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Veszprém
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, San Juan, Puerto Rico
- Slovakia (5):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Martin
  - Novartis Investigative Site, Myjava
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Trnava
- Novartis Investigative Site, Ankara, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- Enalapril: No study treatment (aliskiren or enalapril) was administered in this off-therapy non-interventional second extension study. The arm/group in this second extension study refers to the actual treatment arm/group assigned at the end of the first extension study (Study CSPP100A2365E1: ClinicalTrials.gov Identifier: NCT01151410). During Study CSPP100A2365E1, participants were to receive one of the following doses of enalapril based on their weight: low weight (≥20 to <50 kg) participants - starting dose 2.5 mg with optional titration to 5 and then 10 mg; mid weight (≥50 to <80 kg) participants - starting dose 5 mg with optional titration to 10 and then 20 mg; high weight (≥80 to ≤150 kg) participants - starting dose 10 mg with optional titration to 20 and then 40 mg.
- Aliskiren: No study treatment (aliskiren or enalapril) was administered in this off-therapy non-interventional second extension study. The arm/group in this second extension study refers to the actual treatment arm/group assigned at the end of the first extension study (Study CSPP100A2365E1: ClinicalTrials.gov Identifier: NCT01151410). During Study CSPP100A2365E1, participants were to receive one of the following doses of aliskiren based on their weight: low weight (≥20 to <50 kg) participants - starting dose 37.5 mg with optional titration to 75 and then 150 mg; mid weight (≥50 to <80 kg) participants - starting dose 75 mg with optional titration to 150 and then 300 mg; high weight (≥80 to ≤150 kg) participants - starting dose 150 mg with optional titration to 300 and then 600 mg.
Period: Overall Study
Arm/Group | Enalapril | Aliskiren
Started | 51 | 55
Completed | 49 | 50
Not Completed | 2 | 5
Not completed — Administrative problems | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enalapril | Aliskiren | Total
Number analyzed (Participants) | 51 | 55 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.5 (3.32) | 11.4 (3.21) | 11.4 (3.25)
Age, Customized [Count of Participants; unit: Participants]
  Age group: Children 6 - 11 years | 28 | 30 | 58
  Age group: Adolescents 12 - 17 years | 23 | 25 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 42
  Male | 32 | 32 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 7 | 15
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 30 | 41 | 71
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 14 | 9 | 23
  Ethnicity: Mixed ethnicity | 1 | 3 | 4
  Ethnicity: Other | 36 | 43 | 79
  Ethnicity: Chinese | 0 | 0 | 0
  Ethnicity: Indian (Indian subcontinent) | 0 | 0 | 0
  Ethnicity: Japanese | 0 | 0 | 0
Hypertension etiology [Count of Participants; unit: Participants]
  Primary | 41 | 46 | 87
  Secondary | 10 | 9 | 19
Height [Mean (Standard Deviation); unit: cm] | 151.9 (20.72) | 150.4 (19.31) | 151.1 (19.92)
Weight [Mean (Standard Deviation); unit: kg] | 63.8 (29.99) | 62.6 (30.33) | 63.2 (30.03)
Weight category [Count of Participants; unit: Participants]
  >= 20 kg and < 50 kg | 21 | 24 | 45
  >= 50 kg and < 80 kg | 14 | 17 | 31
  >= 80 kg and <= 150 kg | 16 | 14 | 30
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (7.58) | 26.1 (8.09) | 26.1 (7.81)
BMI category [Count of Participants; unit: Participants]
  < 95th percentile | 49 | 52 | 101
  >= 95th percentile | 2 | 3 | 5
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 104.2 (24.86) | 112.1 (19.39) | 108.3 (22.43)
eGFR category [Count of Participants; unit: Participants]
  < 60 mL/min/1.73m^2 | 1 | 0 | 1
  >= 60 and < 90 mL/min/1.73m^2 | 11 | 5 | 16
  >= 90 mL/min/1.73m^2 | 39 | 50 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight Assessments From Baseline (Visit 2 of the Core Study) to Long Term (LT) Visit 18 (Week 104) for the Enrolled to Follow-up Set (EFS)
Description: Participant weight was measured at Baseline (Visit 2 of the Core study), LT Visit 17, LT Visit 18 ([Week 104] only for participants identified in the core study as having primary hypertension), and LT Visit 19 ([Week 156] only for participants identified in the core study as having secondary hypertension). Body weight was measured to the nearest 0.1 kg in indoor clothing, but without shoes.
Time Frame: Baseline to LT Visit 18 (Week 104): 2 years (104 weeks)
Population: The EFS consisted of all participants who signed the informed consent form (ICF) for the second extension study. Number of participants is the number of EFS participants with non-missing measurement at LT Visit 18. Participants with missing data at LT Visit 18 were not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Enalapril | Aliskiren
Number analyzed (Participants) | 49 | 50
kg | 8.90 (1.359) | 9.22 (1.399)
Statistical Analysis 1: Comparison: Enalapril vs Aliskiren; Test type: Superiority; p = 0.840, ANCOVA — p-value for statistical significance at 0.05 level for 2-sided superiority testing; Treatment regimen, region, age strata, and hypertension etiology (primary, secondary) as factors, and Baseline weight as covariates; Mean Difference (Net) = 0.31, 95% CI 2-sided [-2.74 to 3.37]

2. Primary Outcome: Change in Height Assessments From Baseline (Visit 2 of the Core Study) to Long Term (LT) Visit 18 (Week 104) for the EFS
Description: Participant height was measured at Baseline (Visit 2 of the Core study), LT Visit 17, LT Visit 18 ([Week 104] only for participants identified in the core study as having primary hypertension), and LT Visit 19 ([Week 156] only for participants identified in the core study as having secondary hypertension).
Time Frame: Baseline to LT Visit 18 (Week 104): 2 years (104 weeks)
Population: The EFS consisted of all participants who signed the ICF for the second extension study. Number of participants is the number of EFS participants with non-missing measurement at LT Visit 18. Participants with missing data at LT Visit 18 were not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Enalapril | Aliskiren
Number analyzed (Participants) | 49 | 50
cm | 7.27 (0.586) | 7.96 (0.607)
Statistical Analysis 1: Comparison: Enalapril vs Aliskiren; Test type: Superiority; p = 0.303, ANCOVA — p-value for statistical significance at 0.05 level for 2-sided superiority testing; Treatment regimen, region, age strata, and hypertension etiology (primary, secondary) as factors, and Baseline height as covariates; Mean Difference (Net) = 0.69, 95% CI 2-sided [-0.63 to 2.02]

3. Primary Outcome: Change in BMI Assessments From Baseline (Visit 2 of the Core Study) to Long Term (LT) Visit 18 (Week 104) for the EFS
Description: Participant height and weight was measured at Baseline (Visit 2 of the Core study), LT Visit 17, LT Visit 18 ([Week 104] only for participants identified in the core study as having primary hypertension), and LT Visit 19 ([Week 156] only for participants identified in the core study as having secondary hypertension). BMI was derived.
Time Frame: Baseline to LT Visit 18 (Week 104): 2 years (104 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Enalapril | Aliskiren
Number analyzed (Participants) | 49 | 50
kg/m^2 | 1.53 (0.487) | 1.56 (0.502)
Statistical Analysis 1: Comparison: Enalapril vs Aliskiren; Test type: Superiority; p = 0.957, ANCOVA — p-value for statistical significance at 0.05 level for 2-sided superiority testing; Treatment regimen, region, age strata, and hypertension etiology (primary, secondary) as factors, and Baseline BMI as covariates; Mean Difference (Net) = 0.03, 95% CI 2-sided [-1.06 to 1.12]

4. Primary Outcome: Change in Neurocognitive Assessments From Baseline (Visit 2 of the Core Study) to Long Term (LT) Visit 18 (Week 104) for the EFS
Description: All participants who were determined to have secondary hypertension in the core study and had a Baseline (Visit 2) standardized neurocognitive assessment in the core study received follow-up neurocognitive assessments at LT Visit 18 and LT Visit 19 with the same tool. The neurocognitive assessment of development included assessment of the following abilities: Attention, Processing speed, Working memory, and Motor speed. For Numbers (Forward and Backward Raw Score), Visual Matching (Number Correct), Sequences (Total Raw Score): positive change indicates a numerical increase, which is considered a better outcome/improvement; negative change/numerical decrease is considered a worse outcome/decline. For Visual Matching (Time to Complete), Time Tapping (Right and Left Hands), and Timed Gait: positive change indicates a numerical increase, which is considered a worse outcome/decline; negative change/numerical decrease is considered a better outcome/improvement.
Time Frame: Baseline to LT Visit 18 (Week 104): 2 years (104 weeks)
Population: The EFS consisted of all participants who signed the ICF for the second extension study. Number of participants is those with secondary hypertension and both baseline and LT Visit 18 observations for that test.
Measure: Count of Participants; unit: Participants
Arm/Group | Enalapril | Aliskiren
Number analyzed (Participants) | 8 | 6
Participants
  Numbers: Forward raw score: Positive change | 8 | 4
  Numbers: Forward raw score: No change | 0 | 1
  Numbers: Forward raw score: Negative change | 0 | 1
  Numbers: Backward raw score: Positive change | 5 | 4
  Numbers: Backward raw score: No change | 2 | 1
  Numbers: Backward raw score: Negative change | 1 | 1
  Visual matching: Number correct: Positive change | 7 | 6
  Visual matching: Number correct: No change | 0 | 0
  Visual matching: Number correct: Negative change | 1 | 0
  Visual matching: Time to complete (sec): Positive change | 0 | 0
  Visual matching: Time to complete (sec): No change | 7 | 6
  Visual matching: Time to complete (sec): Negative change | 1 | 0
  Sequences: Total raw score: Positive change | 6 | 6
  Sequences: Total raw score: No change | 1 | 0
  Sequences: Total raw score: Negative change | 1 | 0
  Time tapping: Right hand: Positive change | 7 | 3
  Time tapping: Right hand: No change | 0 | 0
  Time tapping: Right hand: Negative change | 1 | 3
  Time tapping: Left hand: Positive change | 4 | 2
  Time tapping: Left hand: No change | 3 | 2
  Time tapping: Left hand: Negative change | 1 | 2
  Timed gait: Number of seconds: number analyzed (Participants) | 8 | 5
  Timed gait: Number of seconds: Positive change | 4 | 3
  Timed gait: Number of seconds: No change | 3 | 0
  Timed gait: Number of seconds: Negative change | 1 | 2

5. Secondary Outcome: Change in Weight Assessments From Baseline (Visit 2 of the Core Study) to End of Study (EOS) by Hypertension Group
Description: as for outcome 1
Time Frame: Baseline to EOS (2 to 3 years). EOS was defined as LT Visit 18 (Week 104) and LT Visit 19 (Week 156) for participants with primary and secondary hypertension, respectively.
Population: The EFS consisted of all participants who signed the ICF for the second extension study. Number of participants is the number of EFS participants with non-missing measurement at EOS. EOS was defined as LT Visit 18 (Week 104) and LT Visit 19 (Week 156) for participants with primary and secondary hypertension, respectively.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Enalapril | Aliskiren
Number analyzed (Participants) | 41 | 44
kg
  Primary Hypertension Group | 8.31 (1.195) | 8.33 (1.182)
  Secondary Hypertension Group: number analyzed (Participants) | 8 | 7
  Secondary Hypertension Group | -0.73 (3.699) | -3.80 (3.445)
Statistical Analysis 1: Comparison: Enalapril vs Aliskiren; Primary Hypertension group (at LT Visit 18 [Week 104]); Test type: Superiority; p = 0.992, ANCOVA — p-value for statistical significance at 0.05 level for 2-sided superiority testing; Treatment regimen, region, age strata, and Baseline weight as covariates; Mean Difference (Net) = 0.02, 95% CI 2-sided [-3.29 to 3.33]
Statistical Analysis 2: Comparison: Enalapril vs Aliskiren; Secondary hypertension group (at LT Visit 19 [Week 156]); Test type: Superiority; p = 0.215, ANCOVA — p-value for statistical significance at 0.05 level for 2-sided superiority testing; Treatment regimen, region, age strata, and Baseline weight as covariates; Mean Difference (Net) = -3.06, 95% CI 2-sided [-8.22 to 2.10]

6. Secondary Outcome: Change in Height Assessments From Baseline (Visit 2 of the Core Study) to EOS by Hypertension Group
Description: as for outcome 2
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Enalapril | Aliskiren
Number analyzed (Participants) | 41 | 44
cm
  Primary Hypertension Group | 6.80 (0.529) | 7.42 (0.528)
  Secondary Hypertension Group: number analyzed (Participants) | 8 | 7
  Secondary Hypertension Group | 16.05 (3.316) | 16.96 (3.044)
Statistical Analysis 1: Comparison: Enalapril vs Aliskiren; Primary Hypertension group (at LT Visit 18 [Week 104]); Test type: Superiority; p = 0.403, ANCOVA — p-value for statistical significance at 0.05 level for 2-sided superiority testing; Treatment regimen, region, age strata, and Baseline height as covariates; Mean Difference (Net) = 0.62, 95% CI 2-sided [-0.85 to 2.09]
Statistical Analysis 2: Comparison: Enalapril vs Aliskiren; Secondary hypertension group (at LT Visit 19 [Week 156]); Test type: Superiority; p = 0.670, ANCOVA — p-value for statistical significance at 0.05 level for 2-sided superiority testing; Treatment regimen, region, age strata, and Baseline height as covariates; Mean Difference (Net) = 0.92, 95% CI 2-sided [-3.74 to 5.57]

7. Secondary Outcome: Change in BMI Assessments From Baseline (Visit 2 of the Core Study) to EOS by Hypertension Group
Description: Participant weight and height was measured at Baseline (Visit 2 of the Core study), LT Visit 17, LT Visit 18 ([Week 104] only for participants identified in the core study as having primary hypertension), and LT Visit 19 ([Week 156] only for participants identified in the core study as having secondary hypertension). Body weight was measured to the nearest 0.1 kg in indoor clothing, but without shoes. BMI was derived.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Enalapril | Aliskiren
Number analyzed (Participants) | 41 | 44
kg/m^2
  Primary Hypertension Group | 1.30 (0.428) | 1.19 (0.424)
  Secondary Hypertension Group: number analyzed (Participants) | 8 | 7
  Secondary Hypertension Group | -1.81 (1.336) | -2.97 (1.397)
Statistical Analysis 1: Comparison: Enalapril vs Aliskiren; Primary Hypertension group (at LT Visit 18 [Week 104]); Test type: Superiority; p = 0.860, ANCOVA — p-value for statistical significance at 0.05 level for 2-sided superiority testing; Treatment regimen, region, age strata, and Baseline BMI as covariates; Mean Difference (Net) = -0.11, 95% CI 2-sided [-1.29 to 1.08]
Statistical Analysis 2: Comparison: Enalapril vs Aliskiren; Secondary hypertension group (at LT Visit 19 [Week 156]); Test type: Superiority; p = 0.320, ANCOVA — p-value for statistical significance at 0.05 level for 2-sided superiority testing; Treatment regimen, region, age strata, and Baseline BMI as covariates; Mean Difference (Net) = -1.17, 95% CI 2-sided [-3.66 to 1.32]

8. Secondary Outcome: Change in Neurocognitive Assessments From Baseline (Visit 2 of the Core Study) to EOS by Hypertension Group
Description: as for outcome 4
Time Frame: Baseline to EOS (3 years). EOS was defined as LT Visit 19 (Week 156) for participants with secondary hypertension.
Population: The EFS consisted of all participants who signed the ICF for the second extension study. Number of participants is those with secondary hypertension and both baseline and LT Visit 19 observations for that test.
Measure: Count of Participants; unit: Participants
Arm/Group | Enalapril | Aliskiren
Number analyzed (Participants) | 8 | 6
Participants
  Numbers: Forward raw score: Positive change | 7 | 5
  Numbers: Forward raw score: No change | 1 | 0
  Numbers: Forward raw score: Negative change | 0 | 1
  Numbers: Backward raw score: Positive change | 5 | 4
  Numbers: Backward raw score: No change | 2 | 1
  Numbers: Backward raw score: Negative change | 1 | 1
  Visual matching: Number correct: Positive change | 6 | 6
  Visual matching: Number correct: No change | 0 | 0
  Visual matching: Number correct: Negative change | 2 | 0
  Visual matching: Time to complete (sec): Positive change | 0 | 0
  Visual matching: Time to complete (sec): No change | 7 | 6
  Visual matching: Time to complete (sec): Negative change | 1 | 0
  Sequences: Total raw score: Positive change | 8 | 6
  Sequences: Total raw score: No change | 0 | 0
  Sequences: Total raw score: Negative change | 0 | 0
  Time tapping: Right hand: Positive change | 5 | 1
  Time tapping: Right hand: No change | 2 | 1
  Time tapping: Right hand: Negative change | 1 | 4
  Time tapping: Left hand: Positive change | 2 | 2
  Time tapping: Left hand: No change | 3 | 1
  Time tapping: Left hand: Negative change | 3 | 3
  Timed gait: Number of seconds: Positive change | 4 | 3
  Timed gait: Number of seconds: No change | 2 | 0
  Timed gait: Number of seconds: Negative change | 2 | 3

ADVERSE EVENTS:
Time Frame: This study only collected the occurrence of Serious Adverse Events (SAEs) occurring within the first 30 days after the participant had completed the first extension study. SAEs experienced after this 30 day period were reported to Novartis/Noden only if the investigator suspected a causal relationship to the study drug. Every SAE, within the above timeframe was to be reported to Novartis/Noden within 24 hours of learning of its occurrence.
Arm/Group | Enalapril | Aliskiren
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/51 | 0/55
Other Adverse Events (participants affected / at risk) | 0/51 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enalapril (N=51) | Aliskiren (N=55)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0

LIMITATIONS AND CAVEATS:
Due to small sample sizes in the secondary hypertension etiology subgroups, the corresponding p-values for treatment comparisons should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contract with new study sponsor "Noden Pharma".

DOCUMENTS (2):
  • Study Protocol (2011-06-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT01420068/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT01420068/SAP_001.pdf